CLINICAL TRIAL: NCT05262634
Title: Pregnancy Outcome in Women With an Iron Deficiency in the First Trimester
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-02033; bb22Hoesli2
Record Dates: First submitted 2022-02-21; First posted 2022-03-02 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Iron Deficiency
Keywords: iron deficiency anemia of pregnancy; pregnancy outcome; perinatal risk; maternal risk
MeSH Terms: conditions — Iron Deficiencies | interventions — Data Collection; Laboratories

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- study group: iron deficiency: Pregnant women with a documented iron deficiency in the first trimester
  Interventions: Other: Data collection (laboratory and obstetric results)
- control group: normal iron status: Pregnant women with normal hematological parameters and iron status in the first trimester
  Interventions: Other: Data collection (laboratory and obstetric results)

INTERVENTIONS:
Other: Data collection (laboratory and obstetric results) — Maternal data: age, pregnancy, parity, singleton or multiple pregnancy, BMI, obstetric history data, and ethnicity.
  Laboratory chemical results: hemoglobin (Hb), number of erythrocytes, mean corpuscular volume (MCV), mean corpuscular hemoglobin (MCH), number of hypochromic erythrocytes (HRC), erythrocyte distribution width (EBW), ferritin, C reactive protein (CRP).
  Maternal pregnancy outcomes and complications: Hb before and after delivery, mode of delivery, placenta abruption, preeclampsia/eclampsia, gestational diabetes, gestational cholestasis, pregnancy-induced hypertension, bacteriuria or urinary tract infections, peripartum and postpartum hemorrhage, puerperal infections, uterine subinvolution.
  Perinatal outcomes: gestational age, birth weight, intrauterine growth retardation, preterm birth, macrosomia, premature rupture of membranes, Apgar score, intrauterine fetal death, pH values, admission to neonatology

SUMMARY:
The primary aim of this retrospective, monocentric study with two parallel groups is to investigate pregnancy outcome in women with iron deficiency in the first trimester. It compares the pregnancy outcome between pregnant women with an iron deficiency and those without an iron deficiency in the first trimester. The study group are pregnant women with a diagnosed iron deficiency in the first trimester, a total of 227 pregnant women. The control group consists of 486 pregnant women without first-trimester iron deficiency. Matching criteria include parity and maternal age. Data from patient files of pregnant women who were treated in the Women's Clinic, University Hospital Basel between 2017 and 2019 are analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with a documented iron deficiency in the first trimester
* Pregnant women with normal hematological parameters and iron status in the first trimester
* Treated at the Women's Clinic, University Hospital in Basel

Exclusion Criteria:

* Pregnant women with a documented rejection

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The data comes from the patient files of pregnant women who were treated in the Polyclinic Women's Clinic University Hospital Basel between 2017 and 2019.
Sampling Method: Probability Sample
Enrollment: 713 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Proportion of anemia | one time assessment at baseline
  Proportion of anemia in pregnant women with an iron deficiency diagnosed in the first trimester compared to pregnant women with normal hematological parameters and iron status in the first trimester
Proportion of hemorrhage | one time assessment at baseline
  Proportion of hemorrhage in pregnant women with an iron deficiency diagnosed in the first trimester compared to pregnant women with normal hematological parameters and iron status in the first trimester
Proportion of growth retardation | one time assessment at baseline
  Proportion of growth retardation in pregnant women with an iron deficiency diagnosed in the first trimester compared to pregnant women with normal hematological parameters and iron status in the first trimester

CONTACTS AND LOCATIONS:
Overall Officials: Irene Hoesli, Prof. Dr. med., Study Director — Women's Clinic, University Hospital Basel; Gabriela Amstad Bencaiova, Dr. med., Principal Investigator — Women's Clinic, University Hospital Basel
Locations (1):
- Women's Clinic, University Hospital Basel, Basel, Switzerland